CLINICAL TRIAL: NCT03623737
Title: A Randomized Phase II/III Study of Paclitaxel/Cisplatin Versus Cisplatin/5-fluorouracil in Neoadjuvant Chemoradiation Followed by Surgery for Patients With Locally Advanced Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: Comparing Paclitaxel/Cisplatin and Cisplatin/5-fluorouracil in Neo-CRT for ESCC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201606102MIPB
Record Dates: First submitted 2017-06-27; First posted 2018-08-09 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Esophageal Squamous Cell Carcinoma; Chemoradiation
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Neoadjuvant Therapy; Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- paclitaxel plus cisplatin (Experimental): A. T: Paclitaxel 50 mg/m2, 1h IVF, weekly, week 1 to week 5 during CRT. B. P: Cisplatin 30 mg/m2, 2 h IVF, weekly following paclitaxel, week 1 to week 5 during CRT.
  Interventions: Drug: neoadjuvant chemoradiation
- cisplatin plus 5-fluorouracil (Active Comparator): A. P: Cisplatin 75 mg/m2, 2 h IVF, on day 1 of week 1 and week 5 during CRT. B. F: 5-FU 1,000 mg/m2, 24 h IVF, on day 1, 2, 3, 4 of week 1 and week 5 during CRT.
  Interventions: Drug: neoadjuvant chemoradiation

INTERVENTIONS:
Drug: neoadjuvant chemoradiation — Neoadjuvant chemoradiation:
  1. Radiation: 180cGy/fraction, once daily, 5 days a week, to a total of 4,500cGy.
  2. Chemotherapy: Arm A or Arm B Surgery: esophagectomy and 3-fields lymph node dissection
  Other Names: esophagectomy

SUMMARY:
This clinical trial has two stages: phase II and phase III. Eligible patients will be randomized 1:1 to the two arms: paclitaxel plus cisplatin and cisplatin plus 5-fluorouracil. The phase II stage will enroll 128 patients, 64 patients for each arm. The endpoint of the phase II stage is complete pathological response (pCR). If the endpoint, i.e., the significant improvement of pCR rate, is met, the clinical trial will proceed to the phase III stage, in which 120 more patients will be enrolled. The estimated enrollment time is four years with 3 more years of follow-up after completing enrollment. The primary endpoint of the clinical trial is overall survival, and the secondary endpoints include clinical response, disease free survival, operation rate, complete resection rate, tumor regression rate, hospital stay days after surgery, safety and toxicity, and quality of life.

DETAILED DESCRIPTION:
Stage 1: Neoadjuvant chemoradiation (CRT):

Stage 2: Evaluation of clinical responses

1. Evaluation will be done at 3±1 weeks after completing the last fraction of radiotherapy.
2. Evaluation will be performed with panendoscopy, endoscopic ultrasonography (EUS), computed tomography (CT), and positron emission tomography (PET).

Stage 3: Surgery

1. Patients will receive esophagectomy with two field lymph node dissection unless:

   A. Patients become medically unfit for surgery. B. Tumor becomes metastatic or unresectable. C. Patients refuse surgery.
2. Patients who do not receive surgery will go on a second section of CRT:

   A. Radiation: 180cGy/fraction, once daily, 5 days a week, up to a total of 6,300cGy.

   B. Arm A:

   i. T: Paclitaxel 50 mg/m2, 1h IVF, weekly, week 1 to week 3 during CRT. ii. P: Cisplatin 30 mg/m2, 2 h IVF, weekly following paclitaxel, week 1 to week 3 during CRT.

   C. Arm B:

   i. P: Cisplatin 75 mg/m2, 2 h IVF, on day 1 of week 1 during CRT. ii. F: 5-FU 1,000 mg/m2, 24 h IVF, on day 1, 2, 3, 4 of week 1 during CRT.
3. Patients, who receive surgery with R2 resection or the pathology showing positive margins or extracapsular invasion of regional lymph nodes, will also receive the second section of CRT described in above-mentioned stage 3-2.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven squamous cell carcinoma of the intrathoracic esophagus.
2. Locally advanced disease, which is defined by the TNM system of the American Joint Committee on Cancer (AJCC) Cancer Staging System (7th edition), fulfilling one of the following criteria as determined by endoscopic ultrasound, computed tomography, bronchoscopy and positron emission tomography:

   A. T3/4a, N0, M0; B. T1-3, N1-3, M0;
3. Tumor length longitudinal ≤ 8cm and radial ≤ 5cm.
4. The tumor must not extend more than 2cm into the stomach.
5. The tumor must not involve cervical esophagus.
6. No invasion of the tracheobronchial tree or presence of tracheoesophageal fistula.
7. Age ≥ 20 and ≤ 75 years old.
8. Performance status ECOG 0~2.
9. Adequate bone marrow reserves, defined as:

   A. white blood cells (WBC) ≥ 4,000/µl or neutrophil count (ANC) ≥ 2,000/µl; B. platelets ≥ 100,000/µl.
10. Adequate liver function reserves, defined as:

    A. hepatic transaminases ≤ 2.5 x upper limit of normal (ULN); B. serum total bilirubin ≤ 2.0 x upper limit of normal (ULN).
11. Adequate renal function: Creatinine ≤1.5 x upper normal limit or estimated creatinine clearance ≥ 50 ml/min (estimated by Cockcroft-Gault formulation)
12. Written informed consent.
13. Patients must be able to fill in quality of life questionnaires.

Exclusion Criteria:

1. Adenocarcinoma.
2. Previous thoracic irradiation.
3. Previous systemic chemotherapy
4. Synchronously diagnosed squamous cell carcinoma of aerodigestive way, other than esophageal cancer.
5. Prior malignancy, except for the following:

   A. adequately treated basal cell or squamous cell skin cancer; B. in-situ cervical cancer; C. a "cured" malignancy more than 5 years prior to enrollment.
6. Significant co-morbid disease, which prohibits the conduction of chemotherapy, concurrent chemo- radiotherapy, or radical surgery, such as active systemic infection, symptomatic cardiac or pulmonary disease, or psychiatric disorders.
7. Documented myocardial infarction within the 6 months preceding registration (pretreatment ECG evidence of infarct only will not exclude patients). Patients with a history of significant ventricular arrhythmia requiring medication. Patients with a history of 2nd or 3rd degree heart block.
8. Pre-existing motor or sensory neurotoxicity greater than grade 1.
9. Patients with prior allergic reactions to drug containing Cremophor, such as teniposide or cyclosporine.
10. Weight loss > 15%.
11. Dementia or altered mental status that would prohibit the understanding and completion of informed consent and questionnaires.
12. Estimated life expectancy less than 3 months.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
pathological complete response | 2 years
  No cancer cells in primary tumor and all lymph nodes resected are observed by pathologists

SECONDARY OUTCOMES:
Overall survival | 4 years
  Time from enrollment to death
disease free survival | 4 years
  From the day of surgery with R0 resection to recurrence or death of any reasons
clinical response | 2 years
  The clinical response evaluation for the effect of neoadjuvant CRT will be done around 3±1 weeks after completing CRT.
  Evaluation will be performed with panendoscopy, EUS, CT, and PET.
  Clinical responses assessment will include:
  1. Overall clinical response according to RECIST1.1 and Japanese Esophageal Society (JES)
  2. Endoscopic response criteria according to JES
  3. Metabolic response evaluated by PET
operation rate | 2 years
  The ratio of the number of patients who receive surgery over the number of patients enrolled
R0 resection rate | 2 years
  The ratio of the number of patients with surgical R0 resection over the number of patients who receive surgery
tumor regression grade | 2 years
  A 4-tiered tumor regression grading (TRG) system will be used according to the extent of residual carcinoma in the whole tumor area of the esophageal specimen.
  TRG 1: no residual carcinoma. TRG 2: 1%- 10% residual carcinoma. TRG 3: 11%- 50% residual carcinoma. TRG 4: >50% residual carcinoma
The total score of participants of both arms will be analyzed and compared. | 2 years
  By World Health Organization Quality of Life Brief Version (WHOQOL-BREF) Taiwan version (2005), quality of life will be assessed at enrollment, at the end of neoadjuvant CRT, and 3 months after surgery.
  There are 28 subscales in the questionnaire. Each subscale has 5 scores from 1 (the worst) to 5 (the best). The scores of each subscale are summed to be a total score.
Number of participants with treatment-related adverse events as assessed by the NCI Common Toxicity Criteria (CTC) | 2 years
  By the NCI Common Toxicity Criteria (CTC), version 4.0., number of participants with treatment-related adverse events, all grades and grade 3/4, will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No